CLINICAL TRIAL: NCT04072406
Title: A Self-Directed Mindfulness Meditation Intervention in Gynecologic Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Washington University School of Medicine (Other)
Collaborators: Washington University Department of Psychological and Brain Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201905188
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Stage III Gynecologic Cancer; Stage IV Gynecologic Cancer
Keywords: mindfulness; meditation; behavioral treatment
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I: Usual Care (Active Comparator): * Participants assigned to usual care will receive a packet of instructions with information about how to complete weekly surveys via a link that will be emailed to them
  * Participants in both arms will be asked to complete a total of five surveys: baseline, at the end of each of three weeks, and a final survey one month later
  Interventions: Other: Usual care packet
- Arm II: Mindfulness Meditation (Experimental): * Participants will listen to mindfulness meditations daily over the course of three weeks.
  * Participants in both arms will be asked to complete a total of five surveys: baseline, at the end of each of three weeks, and a final survey one month later
  Interventions: Other: Mindfulness meditation

INTERVENTIONS:
Other: Mindfulness meditation — Participants assigned to either condition who do not have a personal electronic device for listening to meditations or completing survey will receive a loaned device from the study team.
  Arms: Arm II: Mindfulness Meditation
Other: Usual care packet — Participants assigned to either condition who do not have a personal electronic device for listening to meditations or completing survey will receive a loaned device from the study team.
  Arms: Arm I: Usual Care

SUMMARY:
The current study examines the effects of a 3-week, at-home mindfulness mediation intervention (MMI) to address psychological and physical distress in patients with gynecologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years old
* Have a diagnosis of Stage III or IV, progressive or recurrent GC (endometrial, ovarian, fallopian tube, primary peritoneal, cervical, vulvar, vaginal, or other)
* Be native English speakers
* Report ≥ 4 on the National Cancer Care Network (NCCN) Distress Thermometer at the time of recruitment;
* Not currently be practicing weekly meditation
* Be willing to create (or already have) an email address
* Have access to internet via a personal electronic device (or be willing to borrow an internet-enabled tablet from the study team).

Exclusion Criteria:

* <18 years old
* Distress Thermometer ratings ≤ 3
* Non-native English speakers
* Individuals with severe depression, and individuals who are having suicidal thoughts.
* Individuals who are also not willing to create an email address for the purpose of the study (or individuals who do not have an email address already)
* Individuals who are currently practicing weekly meditation
* Due to overlap in surveys for other ongoing trials in the Division of Gynecologic Oncology, patients may not be currently enrolled on protocol IRB#: 201511102 (chemoresistance) or IRB# 201804169 (Cytokine-induced depression).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of anxiety as measured by the Hospital Anxiety and Depression Scale (HADS) | From Baseline to week 3
  -On the 14-item Hospital Anxiety and Depression Scale (HADS) symptoms of anxiety (7) and depression (7) are rated on a scale from 0 (less severe) to 3 (more severe).

SECONDARY OUTCOMES:
Change in symptoms of distress as measured by the National Comprehensive Cancer Network Distress Thermometer | From Baseline to week 3
  -Patients rate distress on a scale from 0 (no distress) to 10 (extreme distress).
Change in symptoms of depression as measured by the Hospital Anxiety and Depression Scale (HADS) | From Baseline to week 3
  -On the 14-item Hospital Anxiety and Depression Scale (HADS) symptoms of anxiety (7) and depression (7) are rated on a scale from 0 (less severe) to 3 (more severe).
Change in symptoms of fatigue as measured by the Brief Fatigue Inventory (BFI) | From Baseline to week 3
  -includes 9 items to measure the severity of fatigue-related symptoms on a scale from 0 (no fatigue) to 10 (fatigue as bad as you can imagine). Items include ratings of fatigue at three time points: fatigue when it is at its "worst," fatigue when it is at its "usual" level, and fatigue as it is experienced "now," in the moment.
Change in overall physical symptoms as measured by the Edmonton Symptoms Associated Scale Revised | From Baseline to week 3
  -The Edmonton Symptoms Assessment Scale Revised is a 10-item scale that measures severity of 10 physical and psychological symptoms (e.g., nausea, drowsiness, tiredness, anxiety) on a scale from 0 (e.g., no nausea) to 10 (e.g., worst possible nausea).
Change in emotion regulation as measured by the Emotion Regulation Questionnaire | From Baseline to week 3
  -measures two emotion regulation strategies, cognitive reappraisal and expressive suppression. Respondents rate 10 items about these strategies on a scale from 1 (strongly disagree) to 7 (strongly agree).
Change in coping as measured by the Cognitive Emotion Regulation Questionnaire | From Baseline to week 3
  -Will assess 20 items from four subscales (acceptance, rumination, positive reappraisal, putting into perspective, and self-blame)
Change in mindfulness as measured by the Five-Facet Mindfulness Questionnaire | From Baseline to week 3
  -Assesses observing, describing, acting with awareness, non-judging, and non-reactivity. Participants rate 15 items on a scale from 1 (never or very rarely true) to 5 (very often or always true).
Change in self-compassion as measured by the Sussex-Oxford Compassion for Self Scale | From Baseline to week 3
  -20-item scale that measures overall compassion for the self. The items are divided into five subscales that correspond to the five components of self-compassion. Items are rated from 1 (not at all true) to 5 (always true).
Change in perceived stress as measured by the Perceived Stress Scale | From Baseline to week 3
  -10-item measure of globally perceived stress. The measure invites participants to retrospectively report their feelings and thoughts about various topics during the last month, including "how often [you] have felt upset because of something that happened unexpectedly," "how often [you] have felt that things were going your way," and "how often [you] could not cope with all the things that you had to do." Participants rate each item on a scale of 0 (Never) to 5 (Very Often), and a higher score indicates greater stress.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Carpenter, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu